CLINICAL TRIAL: NCT05053568
Title: Advanced Image Supported Lead Placement in Cardiac Resynchronization Therapy
Brief Title: Image Supported Lead Placement in CRT
Acronym: ADVISE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: CART-Tech B.V. (Unknown); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Health Holland (Other)
Responsible Party: Principal Investigator, M. Meine, Principal Investigator (MD, PhD), UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL73416.041.20; 404460098327 (Other Grant/Funding Number: ZonMW); LSHM191o3-Ho7o (Other Grant/Funding Number: Health-Holland)
Record Dates: First submitted 2021-08-27; First posted 2021-09-22 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
Keywords: Cardiac Resynchronization Therapy; Image-guided therapy; Lead placement; MRI
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Live visualised, fluoroscopy-fused, image-guided, left ventricular lead placement on the basis of avoiding scar and targeting late mechanically activated segments.
  Interventions: Device: CARTBox
- Control group (No Intervention): Empirical standard-of-care left ventricular lead placement, in line with current CRT implantation guidelines with electrical guiding on the basis of Q-LV sense.

INTERVENTIONS:
Device: CARTBox — CARTBox performs analysis of cardiac MRI scans. The result is a treatment file that displays optimal targets for left ventricular lead implantation in CRT. This file will be used as an overlay with live fluoroscopy during the implantation procedure in the intervention group.
  Arms: Intervention group

SUMMARY:
Cardiac resynchronization therapy (CRT) is an established pacemaker therapy for patients with symptomatic chronic heart failure, but is hampered by a non-response rate of 30-40%. Optimising left ventricular (LV) lead placement is the cornerstone of improving treatment. The optimal location for the lead is remote from scar but within segments demonstrating late electromechanical activation. The present study aims to investigate the efficacy and clinical effect of the use of real-time guided lead placement using cardiac MRI and fluoroscopy in a blinded, multicenter, randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure with LV ejection fraction ≤ 35%;
* New York Heart Association class II, III, or IV (ambulatory);
* Optimal medical treatment that is tolerable;
* Left bundle branch block (LBBB) and QRS ≥ 130 ms, OR non-LBBB and QRS ≥ 150 ms.

Exclusion Criteria:

* Pregnancy or lactation;
* Subjects with impaired renal function (severe renal insufficiency, GFR < 30 ml/min/1.73m2);
* Atrial fibrillation or atrial fibrillation during MRI
* Documented allergic reaction to gadolinium;
* Impossibility to undergo an MRI scan;
* Participation in another clinical study that prohibits any procedures other than standard.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Differences in % of patients with succesfull LV lead location | Direct post-CRT
  Lead location, defined as being within, adjacent, or remote from the pre-defined target.

SECONDARY OUTCOMES:
Change in reverse remodelling and volumetric response | 6 months
  Measured as the relative decrease in LV end-systolic volume, indexed to body surface area (LVESVi). Response defined as LVESVi-reduction ≥ 15%.
Change in EQ-5D-5L | 6, 12 and 24 months
  A quality of life questionnaire
Change in Kansas City Cardiomyopathy Questionnaire | 6, 12 and 24 months
  A quality of life questionnaire
Change in CRT response score | 12 months
  A hierarchical clinical endpoints, combining relative LVESVi-decrease, change in New York Heart Association class, and death at 12 month follow-up.
Health Technology Assessment | 24 months
  The value of image-guided lead placement will be investigated in terms of healthcare expenditure revolving heart failure care. This assesment will be based on a previously conducted preliminary economic analysis.

OTHER OUTCOMES:
Difference in total implantation procedure time. | Direct post-CRT
  Compared between both groups. Measured in minutes.
Difference in total fluoroscopy time during procedure. | Direct post-CRT
  Compared between both groups. Measured in minutes.
Difference in total contrast dose used during procedure. | Direct post-CRT
  Compared between both groups. Measured in dose area product.
Difference in change in QRS duration | Direct post-CRT and 6 months
  Compared between groups and according to LV lead location. Measured in ms.
Difference in change in QRSarea | Direct post-CRT and 6 months
  Compared between groups and according to LV lead location. Measured in μVs.
Difference in Q-LV sense | Direct post-CRT
  Compared between groups and according to LV lead location. Measured in ms.
Difference in pacing threshold | Direct post-CRT
  Compared between groups and according to LV lead location. Measured in mV.
Difference in % of patients with disappearance of apical rocking | Direct post-CRT and 6 months
  Compared between groups and according to LV lead location. Option to assess other indices of mechanical recoordination.

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Meine, MD, PhD, Principal Investigator — UMC Utrecht
Locations (7):
- Netherlands (7):
  - Erasmus MC, Rotterdam, South Holland
  - Amsterdam UMC, Amsterdam
  - UMC Groningen, Groningen
  - Maastricht UMC+, Maastricht
  - St. Antonius Nieuwegein, Nieuwegein
  - UMC Utrecht, Utrecht
  - Isala Zwolle, Zwolle

IPD SHARING:
Plan to Share IPD: Yes
Within legal and ethical limits, deidentified individual clinical trial participant-level data (IPD), generated by our research, can be made available. Upon publication, data will be made available upon reasonable request and in agreement with a collaboration agreement. A data sharing and management plan is provided.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Wouters PC, van Slochteren FJ, Tuinenburg AE, Doevendans PA, Cramer MM, Delnoy PHM, van Dijk VF, Meine M. On-screen image-guided lead placement in cardiac resynchronization therapy: Feasibility and outcome in a multicenter setting. Heart Rhythm O2. 2022 Oct 18;4(1):9-17. doi: 10.1016/j.hroo.2022.10.002. eCollection 2023 Jan. PMID 36713038
- [Background] Wouters PC, van Lieshout C, van Dijk VF, Delnoy PH, Doevendans PA, Cramer MJ, Frederix GW, van Slochteren FJ, Meine M. Advanced image-supported lead placement in cardiac resynchronisation therapy: protocol for the multicentre, randomised controlled ADVISE trial and early economic evaluation. BMJ Open. 2021 Oct 25;11(10):e054115. doi: 10.1136/bmjopen-2021-054115. PMID 34697125
- [Background] Gerrits W, Wouters PC, Chiu CSL, Guglielmo M, Cramer MJ, van der Harst P, Vernooy K, van Stipdonk AMW, van Halm VP, van Dijk VF, Ghani A, Maass AH, Yap SC, van Slochteren FJ, Meine M. Optimizing CRT Lead Placement Accuracy With CMR-Guided On-Screen Targeting: A Randomized Controlled Trial (ADVISE-CRT III). JACC Clin Electrophysiol. 2025 Jun;11(6):1293-1305. doi: 10.1016/j.jacep.2025.01.022. Epub 2025 Mar 19. PMID 40117420